CLINICAL TRIAL: NCT06241963
Title: The Efficacy, Safety and Mechanism of High Definition Transcranial Direct Current Stimulation (HD-tDCS) in the Treatment of Refractory Epilepsy
Brief Title: High Definition Transcranial Direct Current Stimulation (HD-tDCS) for Refractory Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AHMU-tDCS-epilepsy
Record Dates: First submitted 2024-01-04; First posted 2024-02-05 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Transcranial Direct Current Stimulation; EEG; Functional Magnetic Resonance Imaging; Refractory Epilepsy; Transcranial Magnetic Stimulation
Keywords: Refractory Epilepsy; Functional Magnetic Resonance Imaging; EEG; Transcranial magnetic stimulation
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Unilateral real High definition transcranial direct current stimulation (Active Comparator): The left electrical stimulation cathode was placed over CP5 with return electrodes placed at FT7, C1, P03 and P9 . The right electrical stimulation cathode was placed over CP6 with return electrodes placed at FT8, C2, PO4 and P10 .
  In the unilateral treatment group, HD-tDCS treatment based on Epileptic discharge is placed on either the left or right side of the brain.Ten 2-mA sessions were applied for 30 minutes,once a day over 10 consecutive workdays.
  Interventions: Device: Active Comparator: Unilateral real High definition transcranial direct current stimulation
- Bilateral real High definition transcranial direct current stimulation (Active Comparator): The left electrical stimulation cathode was placed over CP5 with return electrodes placed at FT7, C1, P03 and P9 . The right electrical stimulation cathode was placed over CP6 with return electrodes placed at FT8, C2, PO4 and P10 .
  In the bilateral treatment group, HD-tDCS treatment was placed on the left and right sides of the brain, at least eight hours apart.. Twenty 2-mA sessions (ramp-up and ramp-down periods of 30 and 30 seconds, respectively) were applied for 30 minutes,twice a day over 10 consecutive workdays.
  Interventions: Device: Active Comparator: Bilateral real High definition transcranial direct current stimulation
- Sham High definition transcranial direct current stimulation (Sham Comparator): The left electrical stimulation cathode was placed over CP5 with return electrodes placed at FT7, C1, P03 and P9 . The right electrical stimulation cathode was placed over CP6 with return electrodes placed at FT8, C2, PO4 and P10.
  The 30 subjects were randomly divided into two groups, 15 receiving bilateral Sham HD-tDCS and 15 receiving unilateral Sham HD-tDCS.
  Sham HD-tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Interventions: Device: Sham Comparator: Sham High definition transcranial direct current stimulation

INTERVENTIONS:
Device: Active Comparator: Unilateral real High definition transcranial direct current stimulation — Improvement of cortical excitability, unilateral stimulation was effective, and no side effects were observed
  Arms: Unilateral real High definition transcranial direct current stimulation
Device: Active Comparator: Bilateral real High definition transcranial direct current stimulation — Improved cortical excitability, the effect was more obvious than unilateral stimulation, the effect lasted longer, and no side effects were observed
  Arms: Bilateral real High definition transcranial direct current stimulation
Device: Sham Comparator: Sham High definition transcranial direct current stimulation — The sham stimulation is mainly used for blank control, control variables, and exclude the interference of other factors
  Arms: Sham High definition transcranial direct current stimulation

SUMMARY:
To observe the clinical effect and safety of transcranial electrical stimulation on patients with refractory epilepsy before and after treatment and analyze its therapeutic mechanism.

DETAILED DESCRIPTION:
All participants underwent a medical evaluation that included physical examination and routine laboratory studies before and after high definition transcranial direct current stimulation (HD-tDCS) treatment.Upon meeting the inclusion criteria and providing informed consent, each participant will complete clinical assessments by a trained investigator and HD-tDCS treatment at Anhui mental health centre.

At least 90 participants were randomized (1:1:1) to receive "bilateral active" ,"Unilateral active" or "Sham" treatment protocol. The left electrical stimulation cathode was placed over CP5 with return electrodes placed at FT7, C1, P03 and P9 . The right electrical stimulation cathode was placed over CP6 with return electrodes placed at FT8, C2, PO4 and P10 .

In the bilateral treatment group, HD-tDCS treatment was placed on the left and right sides of the brain, at least eight hours apart. Twenty 2-mA sessions (ramp-up and ramp-down periods of 30 and 30 seconds, respectively) were applied for 30 minutes,twice a day over 10 consecutive workdays. In the unilateral treatment group, HD-tDCS treatment based on Epileptic discharge is placed on either the left or right side of the brain.Ten 2-mA sessions were applied for 30 minutes,once a day over 10 consecutive workdays.Sham HD-tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.

Before and after the tDCS treatment, the patients had receiving a battery measure of neuropsychological tests, Magnetic resonance imaging scan in multimodalities, VEEG and Resting motor threshold.

The clinical symptom of participants were followed 4 weeks and 12 weeks after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of refractory epilepsy
* Right-handed and aged 18-50 years old and primary school education or above;
* No major neurological or mental illness, no head injury, alcohol dependence or drug dependence;
* During the experiment, the subjects did not smoke, drink, get sick and take psychotropic drugs, and there were no major life events that caused mood changes.

Exclusion Criteria:

* organic brain injury, neurological diseases or serious physical diseases;
* Have a history of substance abuse and drug dependence, or have used antipsychotic drugs in the past three months, and have serious suicidal tendencies;
* There are contraindications for MRI or EEG or transcranial magnetic stimulation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-12 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The changes of Epilepsy diary | Baseline and 10 workdays post-treatment,and follow-up to 1 months and 3 months
  The reduction of seizure frequency in patients with epilepsy will constitute the primary outcome measure to evaluate the efficacy of HD-tDCS, reflecting the improvement of patients' clinical symptoms. Patients and family members are asked to keep an epilepsy diary to record the time, duration, and status of the seizure.

SECONDARY OUTCOMES:
The changes of VEEG | Baseline and 10 workdays post-treatment,and follow-up to 1 months and 3 months
  The number of discharges recorded by VEEG before and after the intervention, as well as the decrease in epileptiform discharge index, were used as indicators to evaluate the improvement of epilepsy symptoms
The changes of resting-state functional connectivity | Baseline and 10 workdays post-treatment,and follow-up to 1 months and 3 months
  the change of resting-state functional connectivity strength between stimulated target and the whole brain areas will be measured by functional MRI and resting-state EEG.
The changes of resting motor threshold(RMT） | Baseline and 10 workdays post-treatment,and follow-up to 1 months and 3 months
  Previous studies have found that the resting movement threshold is an effective measure of cortical excitability in epilepsy patients, and can better predict the therapeutic effect. An elevated resting movement threshold indicates that the treatment is responding.
The changes of glutamate receptor-mediated intracortical facilitation (ICF) | Baseline and 10 workdays post-treatment,and follow-up to 1 months and 3 months
  ICF is a 120% RMT stimulation administered 15 ms after 90% RMT intensity stimulation, glutamate receptor-mediated intracortical promotion
The changes of GABA-A receptor-mediated short septal cortical inhibition (SICI) | Baseline and 10 workdays post-treatment,and follow-up to 1 months and 3 months
  SICI is 120% RMT administered 4 ms after 80% RMT intensity stimulation in response to GABA-A receptor-mediated short-interval cortical inhibition
The changes of GABA-B receptor-mediated long septal cortical inhibition (LICI). | Baseline and 10 workdays post-treatment,and follow-up to 1 months and 3 months
  LICI is 120% RMT administered 150ms after 120% RMT intensity stimulation in response to GABA-A receptor-mediated long-interval cortical inhibition,
The changes of MoCA Score | Baseline and 10 workdays post-treatment,and follow-up to 1 months and 3 months
  MoCA was developed by Nasreddine et al. based on clinical experience and reference to the MMSE cognitive items and scores, and the final version was finalized in November 2004. We adopted a localized version (Mandarin version，includes 2 alternative versions) in line with the Chinese cultural background.A higher score indicates improvement
The changes of Hamilton Depression Rating Scale (HAMD) Score | Baseline and 10 workdays post-treatment,and follow-up to 1 months and 3 months
  The HAMD is a clinic ian-administered depression assessment and consists of 17 items with a total score range from 0 to 54. A higher score indicates a worse outcome.
The changes of Hamilton Anxiety Scale (HAMA) Score | Baseline and 10 workdays post-treatment,and follow-up to 1 months and 3 months
  The HAMA is a 14-item scale to measure the severity of anxiety symptoms, where each item is rated on a scale from 0 to 4. The HAMA total score ranges from 0 to 56, with lower scores indicating less anxiety symptoms.
The changes of Chinese auditory learning test Score | Baseline and 10 workdays post-treatment,and follow-up to 1 months and 3 months
  A group consists of 15 words, read to the subject at a speed of one per second, after reading, let the patient repeat these 15 words, record the number of words spoken correctly, repeat the above behavior five times, start the timer after the end, let the patient recall 15 words after 30 minutes, and calculate the correct number，The more vocabulary is memorized, the better the score
The changes of TMT (Trail Making Test) Score | Baseline and 10 workdays post-treatment,and follow-up to 1 months and 3 months
  The Trail Making Test (TMT) is divided into two parts, part A and part B. Part A requires the subject to connect 25 Numbers on the paper in sequence, and part B requires the subject to connect 25 Numbers of different colors alternately in sequence. The time it takes for the subject to complete all the Numbers is the subject's final score.the shorter the better.
The changes of Face associative memory Score | Baseline and 10 workdays post-treatment,and follow-up to 1 months and 3 months
  The associative memory was estimated using a face-cued word association test. In the face-cued word association test, participants studied 20 human face photographs presented individually in grayscale on a computer screen for 4 s per face. Each photograph displayed a unique common word that the participants read aloud as each face-word pair was shown. The participants were instructed to memorize the word associated with each face. After the face-word pairs were presented, participants were shown the same 20 faces, individually and in a different and randomized order. They were asked to recall the words that were presented with each face. Each face was scored as correct or incorrect. These processes are carried out 2 times in total. The average number of successful answers was defined as the associative memory score.The more faces you remember correctly, the higher your score.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China